



Participant Identification Number for this trial:

## **CONSENT FORM**

Title of Project: What is the scope for low field MRI to replace cone beam computed tomography in dentistry?

Name of Researcher: Dr. Saoirse O'Toole and Dr Jonathan Davies

| | | | Please in | itial box |
|---|---|---|---|---|
| 1. | I confirm that I have read the information sheet dated 14/03/2025 (version 1) for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | | | |
| _ | | • | Aller Control White a few Control | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time | | | |
| | without giving any reason, without my medical care or legal rights being affected. | | | |
| 3. | I understand that I will need to attend a separate hospital site for my magnetic resonance imaging scan. | | | |
| 4. | I understand that I will then need to return for a visit to discuss the results of my scan and | | | |
| | my care may change because of the new information provided by the scan. | | | |
| 5. | I consent that my deidentified data, trial information and questionnaires answered can be sent to academic partners for analysis as part of the trial. | | | |
| 6 | | | | |
| 6. | I understand that relevant sections of my medical notes and data collected during | | | |
| | the study may be looked at by individuals from regulatory authorities or | | | |
| | from the NHS Trust to monitor the study, where it is relevant to my taking part in this research. | | | |
| | I give permission for these individuals to have access to my records. | | | |
| 7. | I agree to take part in the above study. | | | |
| | Name of Participant | <br>Date | Signature | |
| | Name of Person taking consent | Date | Signature | |